CLINICAL TRIAL: NCT06054152
Title: Prediction of Immunotherapy Efficacy Based on Transcriptome of CX3CR1+T Cell in Peripheral Blood
Brief Title: CX3CR1+T Cell Predict Immunotherapy Efficacy
Status: Completed | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chang Chen, Chief Physician, Secretary of the Party Committee, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: CTPI
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: PD-1 inhibitor based immunotherapy — Patients received at least 4 cycles of PD-1 inhibitor-based immune monotherapy or chemoimmunotherapy. PD-1 drug selection should be limited in 4 types of PD-1 inhibitor approved by China FDA and launched in China and Opdivo or Keytruda.

SUMMARY:
This study aimed to evaluate the correlation between the proportion of flow-sorted CX3CR1+T cells in peripheral blood and the CX3CR1+T-specific gene signature and the efficacy of immunotherapy.

DETAILED DESCRIPTION:
The status and abundance of T cells vary across tumor microenvironments (TMEs) may fundamentally influence response to immunotherapy in non-small cell lung cancer. CX3CR1+ CD8+ T cells showed high migration in and were enriched in the blood, whose amplification is strongly associated with response to anti-PD-1 therapy and better survival. However, the prediction performance of CX3CR1+ T features and characteristics has not been fully validated. This study intends to conduct a clinical trial based on CX3CR1+ CD8+T Cell in peripheral blood to verify the association of proportion and specific transcriptome signature of CX3CR1+T Cell in immunotherapy efficacy prediction. With the help of RECIST 1.1 criteria, the investigators evaluate the clinical response after prescribed cycles of treatment to explore the correlation between peripheral blood markers and immunotherapy efficacy. To develop a low cost, robust and accurate prototype prediction model for NSCLC patients who take anti-PD-1 drugs is investigators final translational purpose.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old;
2. Diagnosed as Non-small cell lung cancer by biopsy before treatment;
3. Prepare to receive PD(L)1 inhibitor monotherapy or combined chemotherapy and antivascular drugs;
4. Lesion imaging can be measured and evaluated by RECIST1.1 standard;
5. Life expectancy exceeds 3 months;
6. ECOG score 0-2;
7. The newly IO treated patients did not receive immunotherapy, chemoradiotherapy before participate in the trial;
8. Sign informed consent and be willing to provide 5ml of peripheral blood for research

Exclusion Criteria:

1. Genetic test showed EGFR and ALK mutations;
2. Patients with other co-morbidities that may affect their follow-up and short-term survival;
3. Patients with any history of antitumor therapy;
4. Patients with a history of other systemic tumors;
5. The ineligible participants assessed by the researchers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced non-small cell lung cancer (stage IIIA-IVB) anticipate to receive primary/first-line immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
objective response rate（ORR） | 4 weeks
  Imaging findings of CR, PR, and stable disease (SD) in all subjects evaluated according to RECIST V1.1 after completing 4 cycles of immunotherapy. best overall response (BoR) was evaluated in participants achieving complete and partial response.

SECONDARY OUTCOMES:
progression-free survival (PFS) | 1 year
  progression-free survival (PFS) defined as time from surgery until disease progression or death from any cause
overall survival (OS) | 1 year
  Overall survival (OS) was defined as the time from surgery until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Chang Chen, MD, Ph.D., Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China; Deping Zhao, MD, Ph.D., Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (2):
- China (2):
  - Hunan cancer hospital, Changsha, Hunan
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zheng L, Qin S, Si W, Wang A, Xing B, Gao R, Ren X, Wang L, Wu X, Zhang J, Wu N, Zhang N, Zheng H, Ouyang H, Chen K, Bu Z, Hu X, Ji J, Zhang Z. Pan-cancer single-cell landscape of tumor-infiltrating T cells. Science. 2021 Dec 17;374(6574):abe6474. doi: 10.1126/science.abe6474. Epub 2021 Dec 17. PMID 34914499
- [Background] Williams HN, Kelley J, Folineo D, Williams GC, Hawley CL, Sibiski J. Assessing microbial contamination in clean water dental units and compliance with disinfection protocol. J Am Dent Assoc. 1994 Sep;125(9):1205-11. doi: 10.14219/jada.archive.1994.0164. PMID 7930182
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34914499/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33658501/